CLINICAL TRIAL: NCT04920565
Title: Evalution of the Efficacy and Safety of Hemoperfusion Use With Polymyxin B un Patients With Severe Endotoxemia With Multiple Organ Dysfunction Syndrome After Complicated Operations With Cardiopulmonary Bypass
Brief Title: Efficacy and Safety of Hemoperfusion With Polymyxin B in Septic Shock Associated With Severe Endotoxemia in Cardiac Surgery Patients (РМХ vs SS)
Acronym: РМХ vs SS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Petrovsky National Research Centre of Surgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21021939
Record Dates: First submitted 2021-06-08; First posted 2021-06-10 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Multiple Organ Dysfunction With Severe Endotoxemia
Keywords: test EAA; endotoxemia; hemoperfusion with Polymyxin B; cardiac syrgery
MeSH Terms: conditions — Endotoxemia | interventions — Hemoperfusion

STUDY DESIGN:
Intervention Model Description: In 10 patients meeting three of the following criteria: SOFA ≥5 points, PCT> 2 ng / ml; CRP> 150 ng / ml, vasopressor use, intestinal paresis and / or positive blood culture data - as well as with an EAA level above 0.6, a hemoperfusion procedure with polymyxin B will be performed for 12 hours.
  - with an initial EAA level of more than 0.9, 2 hemoperfusion procedures will be performed with a difference of 12 hours
Masking Description: Using the matching method, a control group of 10 patients (historical randomization without endotoxemia assessment) with multiple organ dysfunction (SOFA ≥5, use of vasopressors) will be formed using the Oxyris universal set for renal replacement therapy for 72 hours.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cardiac surgery patients with multiple organ dysfunction (Experimental): hemoperfusion procedure with polymyxin B will be performed for 12 hours
  Interventions: Device: hemoperfusion with polymyxin B
- cardiac surgery patients (No Intervention): without hemoperfusion with polymyxin B

INTERVENTIONS:
Device: hemoperfusion with polymyxin B — polymyxin B is covalently immobilized on polystyrene strands, selectively removes endotoxin and at the same time there is no leaching of the ligand, immobilization is carried out by electrostatic interaction and Vanderwals force
  Other Names: PMX 20 R
  Arms: cardiac surgery patients with multiple organ dysfunction

SUMMARY:
Sepsis is a state of multiple organ dysfunction caused by a generalized immune-inflammatory response of the body to an infectious agent, with pronounced heterogeneity and interchangeability of clinical and laboratory manifestations. Violation of autoregulation and multiple organ dysfunctions in case of not timely started and / or ineffective therapy lead to the development of multiple organ failure and thanatogenesis in 40-90% of cases. At the moment, there is no standardized approach to the treatment of the entire pool of sepsis patients. Pharmacological effects on receptors for interleukins and endotoxin, antibiotic therapy and immunoprotection do not allow taking the process under complete control. The pathogenesis and clinical diversity of manifestations dictates the need for a personalized approach based on identifying a group of patients with homogeneous characteristics and the course of the process, where one or another technique would have the greatest benefit. The choice of tactics for extracorporeal therapy should be based on early support of organ function and consistent elimination of high concentrations of trigger compounds (endotoxin, other metabolic products of microorganisms and products of cytolysis of a macroorganism), as well as aimed at minimizing the loss of proteins and immune complexes.

The aim of this clinical study was to assess the efficacy and safety of the selective adsorption of endotoxin in patients with severe multiple organ dysfunction after complicated cardiac surgery.

DETAILED DESCRIPTION:
PMX versus SS (polymyxin B versus septic shock) is a single-center, historic, randomized clinical trial to investigate the safety and efficacy of polymyxin B columns (PMX 20R, Toray) in adult patients with severe endotoxemia for the prevention and correction of septic shock after cardiac surgery. All patients must sign an informed consent prior to surgery. The study group will be represented by patients with severe multiple organ dysfunction (SOFA ≥5 points, PCT> 2 ng / ml; CRP> 150 ng / ml, vasopressor use, intestinal paresis and / or positive blood culture data) and endotoxin activity level on the test EAA is higher than 0.6. Patients by outcome will be divided into 2 groups according to the EAA test values: values from 0.6 to 0.89 (group A) and 0.9 and above (group B).

Due to the presence of renal failure in such patients, hemoperfusion will be performed in combination with the oXiris (Baxter) kit on the Prismaflex (Baxter) apparatus (PMX20R - 12 hours; oXiris - 72 hours). The effectiveness of PMX will be assessed based on the decrease in the EAA value below 0.6 12 hours after the end of the hemoperfusion session. If EAA2 is greater than 0.6 PMX will reconnect.

• For patients with a baseline EAA1 value greater than 0.9, PMX reuse is included in the study protocol and performed 12 hours after the first set is turned off. The EAA3 test runs 12 hours after the PMX2 is turned off.

The safety of hemoperfusion will be assessed based on the presence of side effects (progression of signs of hemodynamic impairment) during the procedure.

The control group will consist of 10 patients (historical randomization without endotoxemia assessment) with septic shock with multiple organ dysfunction (SOFA ≥5, use of vasopressors) using the Oxyris universal renal replacement therapy kit for 72 hours. The comparison group will be formed by the matching method.

Additionally, the following will be assessed: the length of stay in the intensive care unit, mortality on the 14th and 28th days after the operation.

It is also planned to assess the dynamics of changes in the immunological status (cellular and humoral immunity) and microbiota metabolism (the level of aromatic microbial metabolites) during hemoperfusion.

ELIGIBILITY:
Inclusion Criteria:

* SOFA +2 points in comparison with the previous assessment; РСТ more than 2 ng / ml; CRP more than 150 ng / ml; norepinephrine infusion; intestinal paresis; positive data of blood culture; ЕАА more than 0,6

Exclusion Criteria:

* bleeding; heparin-induced thrombocytopenia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
endotoxin activity level | 12 hours after the end of the procedure
  frequency of cases of decrease in EAA below 0.6
vasopressor | 6 hours after the start of the procedure
  frequency of discontinuation of vasopressor infusion

SECONDARY OUTCOMES:
mortality | 14 and 28 day
  frequency
SOFA | 24 hours after the end of the procedure
  dynamics on the SOFA scale
IL6/IL10 | 12, 24 hours after the end of the procedure
  ratio

OTHER OUTCOMES:
adverse events | during the procedure
  frequency

CONTACTS AND LOCATIONS:
Overall Officials: MAXIM BABAEV, D.Sc.(medical), Principal Investigator — Petrovsky NRCS
Locations (1):
- Petrovsky National Reasearch Centre of Surgery, Moscow, Russia